CLINICAL TRIAL: NCT00885040
Title: Investigation of Neurofeedback With Real-Time fMRI in Healthy Volunteers and Patients With Hyperkinetic Movement Disorders
Status: Terminated | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 090118; 09-N-0118
Record Dates: First submitted 2009-04-18; First posted 2009-04-21 (Estimated); Last update posted 2019-06-24 (Actual); Status verified 2019-06-20

CONDITIONS: Movement Disorder; Tourette Syndrome; Healthy Volunteer
Keywords: Neurofeedback; Tourette Syndrome; Healthy Volunteer; Movement Disorder; Brain Activity; fMRI; HV
MeSH Terms: conditions — Movement Disorders; Tourette Syndrome

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

* Many people can learn to use feedback about brain activity to modify that activity, but is it not known if people with Tourette syndrome can modify their brain activity.
* Researchers have evidence that certain areas of the brain are involved in causing tics in people with Tourette syndrome. If people with Tourette syndrome can use feedback about brain activity to modify activity in those parts of the brain, they may be able to modify their brain activity to help control the tics.

Objectives:

* To determine if people with and without Tourette syndrome can learn to use thought to control brain activity.
* To test whether people who have Tourette syndrome can learn to control brain activities, possibly helping to control tics.

Eligibility:

* Healthy volunteers ages 18 and older who are right-handed and are willing to not consume caffeine or alcohol for 24 hours before the study visit.
* Patients with Tourette syndrome who have tics that can be observed and studied.
* All participants must be able to undergo magnetic resonance imaging (MRI) scans.

Design:

* Healthy volunteers (two visits to the NIH Clinical Center over a 2- to 4-week period; visit may last up to 3 hours):
* Screening visit, including physical examination and medical history, and a magnetic resonance imaging (MRI) scan if the individual has not had one performed at the National Institutes of Health in the past year.
* Study visit: Functional MRI (fMRI) scan to allow researchers to see if volunteers can learn to control their brain activity during a scan. Volunteers will be asked to complete tasks as directed during the fMRI scan.
* Patients with Tourette syndrome (three or four outpatient visits over a 4- to 6-week period; each visit may last up to 4 hours):
* Screening visit, including physical examination and medical history, and an MRI scan if the individual has not had one performed at the National Institutes of Health in the past year.
* Evaluation visit to ask questions about Tourette symptoms and to have patients complete questionnaires about their tics and their mental health.
* Study visit: fMRI scan to allow researchers to see if patients can learn to control their brain activity during a scan. Patients will be asked to complete tasks as directed during the fMRI scan.
* Final visit: Researchers will ask questions about tic symptoms, have patients complete questionnaires, and perform a brief exam. Afterward, patients will have an fMRI scan similar to the previous one.
* All participants will be paid a small amount of money in compensation for their participation in the study.

DETAILED DESCRIPTION:
Objective:

The objective of this study is to see if healthy volunteers and patients with hyperkinetic movement disorders such as Tic Disorders (TD) including Tourette Syndrome (TS) are able to learn how to alter their brain activity using feedback during functional magnetic resonance imaging (fMRI), and whether such feedback training can lead to improvement in symptoms in TD patients.

Study population:

This study is to be carried out in three phases. In Phase 1 we will study the feedback technique using fMRI with right-handed adult healthy volunteers, in Phase 2 we intend to study if adult patients with TD are also able to learn the feedback technique, and in Phase 3 we intend to study whether feedback training with fMRI leads to improvement in symptoms in TD patients and whether patients were able to retain the ability to alter their brain activity.

Design:

All subjects will have an initial screening visit to consent and assess their eligibility to participate in the current study. All visits are outpatient.

Subjects will have a clinical MRI when required, a series of functional scans, and at least one structural scan for image registration.

Phase 1: Feasibility Studies

Feasibility of fMRI neurofeedback based on activation levels.

Subjects will perform a neurofeedback fMRI visit, where they will attempt at modulating brain activity level based on the observed feedback signal. Task include motor, motor imagery, or mental thoughts. Functional localization of target regions will be done with a motor task or a blink suppression paradigm. Completed.

1. Feasibility of fMRI neurofeedback based on connectivity

   Subjects will perform two fMRI visits, where they will attempt to learn to modulate their own brain connectivity using feedback of connectivity patterns between two motor regions during a real-time fMRI paradigm. Each session will include a performance evaluation. Data acquisition completed.
2. Feasibility of fMRI neurofeedback based on patterns

Subjects will perform one fMRI visit. A blink suppression paradigm will be used to create a personalized model of urge . Using neurofeedback, subjects attempt to modulate the urge pattern. In progress.

Phase 2: Pilot neurofeedback for brain modulation in TD

TD patients will have an evaluation visit, including clinical evaluations, scales and videotaping and an fMRI visit.

In the fMRI visit, the model of urge will be created based on the brain pattern measure before spontaneous tics. Patients will attempt towill be studied to see if they can learn to alter their brain activity to decrease the fitting to the urge model, in a similar way as the healthy volunteers. In progress.

Phase 3: Pilot neurofeedback fMRI for symptoms improvement in TD patients

TD patients will have one evaluation, one scanning, and one follow-up) visit. No visit will last more than 4 hours. The effect of altering brain activity in a specific brain area on symptoms in TD patients will be studied. Patients will be asked to continue to focus their thoughts as they did during feedback scanning any time that they feel an urge prior to a tic or every hour while awake, whichever is more frequent, until a follow-up visit and fMRI scan two or three days later. Require power analysis based on Phase 2.

Outcome measures:

Primary outcomes

Phase 1

1. The difference in connectivity between two ROIs after feedback training compared to a baseline.
2. The difference in neural pattern after feedback training compared to a baseline.

Phase 2

The difference in neural pattern after feedback training compared to a baseline.

Phase 3

The difference in symptoms measured by a TS rating scale before fMRI scanning compared to two or three days after learning the feedback technique.

Secondary outcomes

Phase 1

1. Changes in motor performance on grooved pegboard test
2. Changes in number of blinks after a successful neurofeedback run.

Phase 2 and 3

Changes in number of tics after successful neurofeedback runs compared to baseline.

ELIGIBILITY:
* INCLUSION CRITERIA:

Healthy Volunteers

1. Aged 18 to 60
2. Right-hand dominant
3. Have a normal neurological exam
4. Have the capacity to give informed consent
5. Willing to abstain from caffeine and alcohol for 24 hours prior to MRI scanning

TD Patients

1. Aged 18 to 60
2. Right-dominant
3. Have TS or chronic motor or vocal tic disorder diagnosis based on neurological examination and meeting criteria of the Diagnostic and Statistical Manual of Mental Disorders 4th 5th Edition (DSM-V)
4. Have the capacity to give informed consent
5. A Yale Global Tic Severity Scale (YGTSS) total score of at least 5
6. Willing to abstain from caffeine and alcohol for 24 hours prior to MRI scanning
7. If pharmacologically treated for TD, willing to not alter medication dosages or regimens between the screening visit and scanning visit for participants of Phase 2 or between the screening visit and follow-up visit for participants of Phase 3

EXCLUSION CRITERIA:

Healthy Volunteers

1. Pregnancy
2. Any abnormal findings on neurological exam
3. Any finding on the MRI safety questionnaire that prevents them from safely undergoing an MRI scan
4. Any medical condition that would prevent them from lying flat for up to 3 hours
5. Any history of central nervous system infection or inflammation, brain tumor, stroke, head trauma or a vascular malformation as obtained by history or from imaging studies
6. Presence of any active or medically treated neurological conditions such as epilepsy, multiple sclerosis, or a movement disorder
7. Presence of any active or medically treated psychiatric problems such as depression, OCD or ADHD
8. Presence of uncontrolled medical illnesses such as heart, lung, or kidney disease
9. Presence of claustrophobia or other restriction that prevents them from undergoing a scan in a confined space for up to 3 hours
10. Presence of continuous or excessive movements at rest or are unable to remain supine while undergoing a scan for up to 3 hours.

TD Patients

1. Pregnancy
2. Any finding on the MRI safety questionnaire that prevents them from safely undergoing an MRI scan
3. Any medical condition that would prevent them from lying flat for up to 3 hours
4. Any history of central nervous system infection or inflammation, brain tumor, stroke, head trauma or a vascular malformation as obtained by history or from imaging studies
5. Presence of uncontrolled psychiatric problems such as depression, OCD or ADHD
6. Patients with a history of a psychotic disorder such as schizophrenia
7. Patients with other movement disorders or progressive neurological disorders other than Tic disorders such as Multiple Sclerosis or epilepsy
8. Presence of uncontrolled medical illnesses such as heart, lung, or kidney disease
9. Presence of claustrophobia or other restrictions that prevent them from undergoing a scan in a confined space for up to 3 hours
10. Presence of continuous or excessive movements at rest or are unable remain supine while undergoing a scan for up to 3 hours
11. Presence of secondary form of tic disorder

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2009-04-17; Study Completion 2019-06-20

PRIMARY OUTCOMES:
Phase 1 & 2: Difference in BOLD signal in a ROI during neurofeedback after training compared to resting baseline. Phase 3: Change in YGTSS measured prior to neurofeedback training compared to the score measured at a follow-up visit.

SECONDARY OUTCOMES:
Difference in BOLD signal in a ROI during neurofeedback compared to a resting baseline after subsequent scanning runs and during a transfer task, and in Phase 3 compared to controls. Also any changes of neurofeedback on various disease measures...

CONTACTS AND LOCATIONS:
Overall Officials: Silvina G Horovitz, Ph.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Albin RL, Mink JW. Recent advances in Tourette syndrome research. Trends Neurosci. 2006 Mar;29(3):175-82. doi: 10.1016/j.tins.2006.01.001. Epub 2006 Jan 23. PMID 16430974
- [Background] Banzett RB, Mulnier HE, Murphy K, Rosen SD, Wise RJ, Adams L. Breathlessness in humans activates insular cortex. Neuroreport. 2000 Jul 14;11(10):2117-20. doi: 10.1097/00001756-200007140-00012. PMID 10923655
- [Background] Baym CL, Corbett BA, Wright SB, Bunge SA. Neural correlates of tic severity and cognitive control in children with Tourette syndrome. Brain. 2008 Jan;131(Pt 1):165-79. doi: 10.1093/brain/awm278. Epub 2007 Dec 3. PMID 18056159